CLINICAL TRIAL: NCT05958381
Title: Treatment of Cognitive Deficits in Multiple Sclerosis With High-Definition Transcranial Direct Current Stimulation
Acronym: MS-HDtDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-521; HT94252310618 (Other Grant/Funding Number: CDMP - MS220175); E04675.1a (Other: OHRO)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: transcranial direct current stimulation (tDCS); multiple sclerosis; electroencephalography (EEG)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 treatment arms: (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 15 sessions to (2) sham tDCS following the same schedule.
  Additionally, after completing the initial active or sham treatment and immediate and 2-month follow-up testing sessions, selected participants will be invited back for newly assigned treatment conditions, 20 minutes over 15 sessions and will be and re-evaluated at immediate- and 2-months follow-up testing sessions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, assessors, and technicians interacting with participants will be blind to assigned conditions. The software for the transcranial direct current system allows for maintaining blinds when uploading and running protocols.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial direct current stimulation (Experimental): Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. Stimulation will consist of 1 milliamp stimulation, with anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.
  Other Names:
  tDCS
  1 milliamp tDCS High definition tDCS High definition transcranial direct current stimulator, Neuroelectrics Starstim tES, SN E20200930-10
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Sham transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. The sham setup will consist of anodal electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, ramp down to 0 milliamps over 60 seconds and then be left off for 20 minutes.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. Stimulation will consist of 1 milliamp stimulation, with anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.
  Other Names: tDCS
  Arms: Transcranial direct current stimulation
Device: Sham transcranial direct current stimulation — Sham transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. The sham setup will consist of anodal electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, ramp down to 0 milliamps over 60 seconds and then be left off for 20 minutes.
  Other Names: Sham tDCS
  Arms: Sham transcranial direct current stimulation

SUMMARY:
The purpose of the study is to test whether low level electric stimulation, called transcranial Direct Current Stimulation (tDCS), on the part of the brain (i.e., presupplementary motor area) thought to aid in memory will improve verbal retrieval in multiple sclerosis patients. The primary outcome measures are neuropsychological assessments of verbal retrieval, and the secondary measures are neuropsychological assessments of other cognitive abilities and electroencephalography (EEG) measures. Additionally, the study will examine the degree to which baseline assessments of cognition and concussion history predict responses to treatment over time, both on assessments administered within the intervention period and at follow-up.

DETAILED DESCRIPTION:
Using two treatment arms, the study will examine improvement of verbal retrieval and other cognitive deficits associated with multiple sclerosis by comparing (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 10 sessions to (2) sham tDCS following the same schedule. Additionally, after completing the initial active or sham treatment and immediate and 2-month follow-up testing sessions, selected participants will be invited back for newly assigned treatment conditions, 20 minutes over 10 sessions and will be re-evaluated at immediate and 2-month follow-up testing sessions.

Patients with multiple sclerosis and observed cognitive deficits will be randomly assigned to one of the two treatment arms (and re-assigned for the second round of intervention, as described above). Primary outcome verbal retrieval measures, secondary neuropsychological and electroencephalography (EEG) measures, and prescreening assessments for study concussion history and contraindications for treatment will be collected prior to being assigned to a treatment arm (i.e., baseline).

Primary outcome verbal retrieval measures and secondary neuropsychological and electroencephalography (EEG) measures will be at baseline and two times following treatment competition (i.e., immediate and 2-months). For participants selected for the second round of intervention, primary outcome verbal memory measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected again two times immediately following completion of the last treatment and 2-months afterward.

ELIGIBILITY:
Inclusion Criteria:

º Diagnosed with relapsing-remitting multiple sclerosis (RRMS)

º Memory retrieval deficit based on neuropsychological testing done in our lab

º Must be fluent in speaking and reading English.

Exclusion Criteria:

º Relapse or acute MS exacerbation or a course of steroids in the two months preceding the testing

º Participants using benzodiazepines must have been on a stable dose for at least two months

º Potentially confounding psychological or neurological disorder, including:

* dementia of any type
* epilepsy or other seizure disorders
* severe traumatic brain injury
* brain tumor
* present drug abuse
* stroke
* blood vessel abnormalities in the brain
* Parkinson's disease
* Huntington's disease

º inability to give informed consent

º cranial implants

º skull defects that affect tDCS administration

º use of medications that interact with or potentially interact with tDCS effects, including:

* anti-convulsants
* L-dopa
* carbamazepine
* sulpiride
* pergolide
* lorazepam
* rivastigmine
* dextromethorphan
* D-cycloserine
* flunarizine
* ropinirole
* stimulants (dextroamphetamine/amphetamine/modafinil/armodafinil) must be stopped during enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment group differences in change from Baseline to 1-week Post-Treatment on Category Fluency | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on Category Fluency from baseline to 1-week post-treatment.
  Metric: Number of Correct Items Generated
Treatment group differences in change from Baseline to 2-months Post-Treatment on Category Fluency | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on Category Fluency from baseline to 2-months post-treatment.
  Metric: Number of Correct Items Generated
Treatment group differences in change from Baseline to 1-week Post-Treatment on COWAT | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on COWAT from baseline to 1-week post-treatment.
  Metric: Number of Correct Items Generated
Treatment group differences in change from Baseline to 2-months Post-Treatment on COWAT | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on COWAT from baseline to 2-months post-treatment.
  Metric: Number of Correct Items Generated

SECONDARY OUTCOMES:
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Trail Making Test (Part A) | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part A) from baseline to 1-week post-treatment.
  Metric: Time to Solution
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Trail Making Test (Part B) | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part B) from baseline to 1-week post-treatment.
  Metric: Time to Solution
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Delis Kaplan Color Word Interference Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Delis Kaplan Color Word Interference Test from baseline to 1-week post-treatment.
  Metric: Time to Name Items
Treatment group differences in change from Baseline to 1-week Post-Treatment on on the Digit Span Forward | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the on the Digit Span Forward from baseline to 1-week post treatment.
  Metric: Memory Span
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Digit Span Backward | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Digit Span Backward from baseline to 1-week post treatment.
  Metric: Memory Span
Treatment group differences in change from Baseline to 1-week Post-Treatment on on the the Rey-Osterrieth Complex Figure Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Rey-Osterrieth Complex Figure Test from baseline to 1-week post treatment.
  Metric: Score
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Digit Symbol Substitution Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the on the the Digit Symbol Substitution Test from baseline to 1-week post treatment.
  Metric: Number of Items
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Grooved Pegboard Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Grooved Pegboard Test from baseline to 1-week post-treatment.
  Metric: Completion Time
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Semantic Object Retrieval Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Object Retrieval Test from baseline to 1-week post-treatment.
  Metric: Number of Correct Names Retrieved
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Boston Naming Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Boston Naming Test from baseline to 1-week post-treatment.
  Metric: Number of Items Correctly Named
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Auditory Verbal Learning Test | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Auditory Verbal Learning Test from baseline to 1-week post-treatment.
  Metric: Number of Items Remembered
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Trail Making Test (Part A) | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part A) from baseline to 2-months post-treatment.
  Metric: Time to Solution
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Trail Making Test (Part B) | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part B) from baseline to 2-months post-treatment.
  Metric: Time to Solution
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Delis Kaplan Color Word Interference Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Delis Kaplan Color Word Interference Test from baseline to 2-months post-treatment.
  Metric: Time to Name Items
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Digit Span Forward | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the on the Digit Span Forward from baseline to 2-months post-treatment.
  Metric: Memory Span
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Digit Span Backward | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the on the Digit Span Backward from baseline to 2-months post-treatment.
  Metric: Memory Span
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Rey-Osterrieth Complex Figure Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the on the Rey-Osterrieth Complex Figure Test from baseline to 2-months post-treatment.
  Metric: Score
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Digit Symbol Substitution Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the on the the Digit Symbol Substitution Test from baseline to 2-months post treatment.
  Metric: Number of Items
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Grooved Pegboard Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Grooved Pegboard Test from baseline to 2-months post-treatment.
  Metric: Completion Time
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Semantic Object Retrieval Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Object Retrieval Test from baseline to 2-months post-treatment.
  Metric: Number of Correct Names Retrieved
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Boston Naming Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Boston Naming Test from baseline to 2-months post-treatment.
  Metric: Number of Items Correctly Named
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Auditory Verbal Learning Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Auditory Verbal Learning Test from baseline to 2-months post-treatment.
  Metric: Number of Items Remembered
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Semantic Inhibition Task EEG spectral power | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Inhibition Task EEG from baseline to 1-week post-treatment.
  Metric: EEG spectral (theta) power
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Semantic Inhibition Task EEG spectral power | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Inhibition Task EEG from baseline to 2-months post-treatment.
  Metric: EEG spectral (theta) power
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Semantic Inhibition Task EEG Event-Related Potential (N2/P3) | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Inhibition Task EEG from baseline to 1-week post-treatment.
  Metric: EEG N2/P3 event-related potential amplitude
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Semantic Inhibition Task EEG Event-Related Potential (N2/P3) | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Inhibition Task EEG from baseline to 2-months post-treatment.
  Metric: EEG N2/P3 event-related potential amplitude
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Semantic Object Retrieval EEG spectral power | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Object Retrieval EEG from baseline to 1-week post-treatment.
  Metric: EEG spectral (theta) power
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Semantic Object Retrieval EEG spectral power | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Object Retrieval EEG from baseline to 2-months post-treatment.
  Metric: EEG event-related potential amplitude
Treatment group differences in change from Baseline to 1-week Post-Treatment on the Semantic Object Retrieval EEG event-related potential | Outcome measures will be assessed as change over a period of 6 weeks: Change from baseline to 1-week Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Object Retrieval EEG from baseline to 1-week post-treatment.
  Metric: EEG late-onset (750 ms) event-related potential
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Semantic Object Retrieval EEG event-related potential | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-months Post-Treatment
  Evaluation of treatment group differences in change on the Semantic Object Retrieval EEG from baseline to 2-months post-treatment.
  Metric: EEG late-onset (750 ms) event-related potential

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, Jr, MD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas at Dallas, Richardson, Texas, United States